CLINICAL TRIAL: NCT01386502
Title: Phase I Trial of Escalating Doses of Anti-PD1 Monoclonal Antibody (CT-011) in Combination With p53 Vaccine in Adults With Advanced Solid Tumors
Brief Title: CT-011 and p53 Genetic Vaccine for Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110198; 11-C-0198
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Breast Cancer; Colon Cancer; Pancreatic Cancer; Sarcoma; Ovarian Cancer
Keywords: Solid Tumors; Monoclonal Antibody; Peptide Vaccine; Toxicity; PD-1 ligand; Solid Tumor; Breast Cancer; Ovarian Cancer; Pancreatic Cancer; Colon Cancer; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Pancreatic Neoplasms; Sarcoma; Ovarian Neoplasms | interventions — p53 peptide 264-272, human; pidilizumab

INTERVENTIONS:
Biological: p53: 264-272 peptide
Drug: CT-011

SUMMARY:
Background:

* The p53 gene normally helps to stop cancer cells from growing. However, when the p53 gene is mutated or damaged, cancer cells may grow unchecked. Researchers have been working on a vaccine that will help the immune system recognize and destroy cells that have the p53 mutation and may be cancerous.
* CT-011 is another drug that may help the body's immune system to fight cancer. This drug blocks a chemical found on tumor cells that prevents the immune system from recognizing and destroying them. Research studies have shown that CT-011 slows the growth of tumors. By combining the p53 vaccine and CT-011, researchers hope to slow or stop tumor growth in people whose cancer that has not responded to standard treatments.

Objectives:

- To test the safety and effectiveness of CT-011 and the p53 genetic vaccine to treat adults with solid tumors that have not responded to standard treatments.

Eligibility:

- People at least 18 years of age who have solid tumors that have not responded to standard treatments.

Design:

* Participants will be screened with a medical history and physical exam. They will also have blood tests and tumor imaging studies.
* Participants will receive the p53 vaccine as an injection in the arm or thigh.
* Two days after receiving the p53 vaccine, those in the study will receive CT-011 as an infusion over about 2 hours. Participants will be monitored during the infusion for any side effects.
* The combination of p53 vaccine and CT-011 will be repeated every 3 weeks (one cycle). Treatment will continue as long as the side effects are not severe and the tumor does not grow.
* Three weeks after the second dose of p53 vaccine and CT-011, participants will have a full physical exam. They will also have blood tests, and tumor imaging studies. This exam set will be repeated after every two cycles of p53 vaccine and CT-011.
* Participants will have regular follow-up visits for up to a year after stopping treatment.

DETAILED DESCRIPTION:
Background:

* PD1 is an inhibitory receptor that belongs to CD28-B7 family.
* PD1 binds to two ligands PD-L1 and PD-L2 to down modulate T-cell immune responses.
* PD1 is expressed on T cells, B cells, and NK cells.
* The over expression of PD-1 ligand (PD-L1) in tumors is associated with an immune suppression and poor prognosis.

Objectives:

* To determine the safety and tolerability of escalating doses of anti PD1 antibody (CT-011) in combination with subcutaneous p53 vaccine.
* To determine the immune response to wt p53 (264-272) peptide.
* To determine the clinical efficacy of this combination.

Eligibility:

* 18 years of age or older, not pregnant or nursing and not immunocompromised or having an autoimmune disease.
* HLA-A2 haplotype.
* ECOG performance status of 0-1.
* Advanced solid tumors over expressing p53 protein with a histological confirmation of the original primary tumor via the Pathology Laboratory, CCR , NCI.

Design:

* Single arm, pilot/phase I trial in patients receiving a fixed dose of vaccine in combination with an escalating dose of CT-011.
* The vaccine will be administered subcutaneously every 3 weeks followed by CT-011 two days after each vaccine until disease progression or toxicity.
* Patients will undergo blood draw or aphaeresis for immunologic assays prior to starting treatment and after every second cycle.
* Patients will be assessed for overall safety, immunologic efficacy, tumor response using RECIST criteria and survival.
* Patients will be followed for up to two years after the last vaccination for assessment of safety and efficacy.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Solid malignancies with a histological confirmation of the original primary tumor via the pathology report for which no curative therapies are available.
  2. Patients must have disease progression after at least one prior first line disease-appropriate therapy, or be unable to tolerate or declined to receive first line therapy.
  3. No chemotherapy or radiation therapy or systemic steroids for at least 4 weeks prior to starting vaccination. No immunotherapy (including monoclonal antibodies) within 4 weeks prior to start of vaccine. Patients should have recovered from all acute toxicities of previous treatment (excluding alopecia).
  4. Patients must have tumors over expressing p53 protein as assessed by immunohistochemistry, as determined by positive staining of tumor sample when compared to negative controls. The immunohistochemical staining will be performed in the Pathology Laboratory, CCR, NCI on fresh or archival tissue and will be supervised by Dr. Merino. The criteria used to determine overexpression will be that used in the Pathology Laboratory: Ten fields will be evaluated at 40 times magnification and if > 25% of cells stain positive, the tumor will be categorized as an overexpressor. Fresh tissue from a new biopsy will only be collected for IHC staining if the tumor is easily accessible and does not pose greater than minimal risk. A separate procedure consent will be required for all biopsy procedures.
  5. Patients must be 18 years of age or older.
  6. Life expectancy of greater than 3 months.
  7. ECOG performance status of 0-1.
  8. ECG with no evidence of arrhythmia, conduction abnormality or ischemia.
  9. Patients must have organ and marrow function as defined below:

     i. Leukocytes greater than or equal to 2,500/mcL

     ii. Lymphocytes greater than or equal to 800/mcL

     iii. ANC greater than or equal to 1000/mcL

     iv. Platelets greater than or equal to 100,000/mcL

     v. Total Bilirubin less than or equal 2mg/dL

     vi. AST (SGOT)/ALT (SGPT) less than or equal to 1.5 times the institutional upper limit of normal (ULN)

     vii. Creatinine less than or equal to 2mg/dL
  10. Patients must have HLA-A0201.
  11. Patients must be willing to travel to the NIH Clinical Center for treatment and follow up visits.
  12. Willing to use effective birth control measures: Since the effects of P53 vaccine and CT-011 on the developing human fetus are unknown and potentially harmful, women of child-bearing potential and men with partners of childbearing potential must agree to use adequate contraception (hormonal or double barrier method of birth control or complete abstinence) prior to study entry and for the duration of study participation and for one month after the last dose of investigational agent. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  13. Patients must understand and sign an informed consent document that explains the neoplastic nature of his/her disease, the procedures to be followed, the experimental nature of the treatment, alternative treatments, and potential risks and toxicities.

EXCLUSION CRITERIA:

1. Concurrent therapy with any other investigational agent(s).
2. Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and frequent development of progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events. Patients with treated brain metastases which have been stable for 6 months or longer will be eligible.
3. Patients who are immunocompromised (HIV positive) or with active Hepatitis B or C; HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with CT-011 or p53. .
4. Patients who have underlying immune deficiency or history of autoimmune disease (including but not limited to SLE, rheumatoid arthritis, multiple sclerosis, inflammatory bowel disease, regional enteritis or other diseases known or presumed to be of autoimmune origin.)
5. Patients being chronically treated with immunosuppressive drugs such as cyclosporin, adrenocorticotropic hormone (ACTH).
6. Concurrent use of systemic steroids except physiologic doses for systemic steroid replacement or local therapy. Physiologic doses are defined as daily systemic therapy used to replace endogenous steroids because of HPA axis dysfunction or other physiological abnormality.
7. History of a second active malignancy in the last 2 years other than non-melanoma skin cancers or carcinoma in situ of the cervix.
8. Patients with active infections requiring antibiotics.
9. Patients with New York Heart Association stage 2 or greater heart failure, unstable angina or cardiac arrhythmias requiring therapy including atrial fibrillation.
10. Pregnant women or nursing mothers are ineligible since the effect of this investigational treatment on the health of the fetus is not known.
11. If, in the opinion of the Principal or Associate Investigators, it is not in the best medical interest of the patient to enter this study, the patient will not be eligible.
12. Patients with history of chronic radiation injury/inflammation due to the risk of perforation in the event of autoimmune inflammation, or history of chronic diarrhea due to previous treatments or surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06-15; Study Completion 2011-10-31 (Actual)

PRIMARY OUTCOMES:
To determine the safety and tolerability of escalating doses of anti PD1 antibody (CT-011) in combination with subcutaneous p53 vaccine.

SECONDARY OUTCOMES:
To determine the immune response to wt p53 (264-272) peptide.
To determine the clinical efficacy of this combination.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ghebeh H, Mohammed S, Al-Omair A, Qattan A, Lehe C, Al-Qudaihi G, Elkum N, Alshabanah M, Bin Amer S, Tulbah A, Ajarim D, Al-Tweigeri T, Dermime S. The B7-H1 (PD-L1) T lymphocyte-inhibitory molecule is expressed in breast cancer patients with infiltrating ductal carcinoma: correlation with important high-risk prognostic factors. Neoplasia. 2006 Mar;8(3):190-8. doi: 10.1593/neo.05733. PMID 16611412
- [Background] Thompson RH, Kuntz SM, Leibovich BC, Dong H, Lohse CM, Webster WS, Sengupta S, Frank I, Parker AS, Zincke H, Blute ML, Sebo TJ, Cheville JC, Kwon ED. Tumor B7-H1 is associated with poor prognosis in renal cell carcinoma patients with long-term follow-up. Cancer Res. 2006 Apr 1;66(7):3381-5. doi: 10.1158/0008-5472.CAN-05-4303. PMID 16585157
- [Background] Hamanishi J, Mandai M, Iwasaki M, Okazaki T, Tanaka Y, Yamaguchi K, Higuchi T, Yagi H, Takakura K, Minato N, Honjo T, Fujii S. Programmed cell death 1 ligand 1 and tumor-infiltrating CD8+ T lymphocytes are prognostic factors of human ovarian cancer. Proc Natl Acad Sci U S A. 2007 Feb 27;104(9):3360-5. doi: 10.1073/pnas.0611533104. Epub 2007 Feb 21. PMID 17360651